CLINICAL TRIAL: NCT04005781
Title: The Effect of Hydroxychloroquine Sulphate on Hedonic Food Intake, Appetite-related Sensations and Gastrointestinal Hormone Release in Overweight Female Subjects
Brief Title: Effect of Bitter in Overweight Female Volunteers
Acronym: PLAQOW
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: S62007
Record Dates: First submitted 2019-06-11; First posted 2019-07-02 (Actual); Last update posted 2019-07-02 (Actual); Status verified 2019-07

CONDITIONS: Obesity
Keywords: bitter; quinine; ghrelin; motilin; food intake
MeSH Terms: conditions — Obesity | interventions — Hydroxychloroquine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hydroxychloroquine sulphate (Experimental): Plaquenil (hydroxychloroquine sulphate) will be acutely administered per os with 240 ml of water. Two tablets of 200 mg hydroxychloroquine sulphate each will be given.
  Interventions: Drug: Hydroxychloroquine sulphate
- Placebo (Placebo Comparator): Two placebo tablets will be acutely administered per os with 240 ml of water.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Hydroxychloroquine sulphate — After a stabilization period of 20 min and 10 min after the first blood collection, Plaquenil (Hydroxychloroquine sulfate) will be administered per os (total dose of 400 mg) in a randomized, double-blinded fashion.
  Other Names: Plaquenil
  Arms: Hydroxychloroquine sulphate
Drug: Placebo — After a stabilization period of 20 min and 10 min after the first blood collection, Placebo will be administered per os (2 tablets) in a randomized, double-blinded fashion.
  Arms: Placebo

SUMMARY:
We want to investigate whether an acute administration of hydroxychloroquine sulphate affects hedonic food intake, appetite related sensations and gastrointestinal hormone release in overweight female subjects.

DETAILED DESCRIPTION:
Intragastric administration of a quinine-solution has shown to decrease hedonic food intake in healthy female volunteers. The effect of a tablet containing hydroxychloroquine sulphate on hedonic food intake in overweight female individuals has not been studied to date. The primary outcome of the current study is to evaluate the effect of hydroxychloroquine sulphate on hedonic food intake, assessed by ad libitum food intake of a chocolate milkshake one hour after dosing. The study is a randomized, placebo-controlled, double blinded cross-over study. Forty overweight females will be recruited. An acute dose of 400 mg hydroxychloroquine sulphate will be administered. Blood samples will be collected at regular time points to measure gastrointestinal hormone release and whole blood glucose levels. Appetite-related sensations will be scored at regular time points on visual analog scales.

ELIGIBILITY:
Inclusion Criteria:

* Subject is female between 18 and 65 years of age.
* Subject has a BMI between 25 and 30 kg/m² and has a stable body weight for at least 3 consecutive months at the start of the study and keeps a stable weight during the study visits.
* Subject is allowed to take 2 Plaquenil capsuls for one visit with a maximal dose of 6.5 mg hydroxychloroquine sulphate per kg bodyweight.
* Women of child-bearing potential agree to apply during the entire duration of the trial a highly effective method of birth control, which is defined as those which result in a low failure rate (i.e., less than 1% per year) when used constantly and correctly such as implants, injectables, combined oral contraceptive method, or some intrauterine devices (IUDs), sexual abstinence, or vasectomized partner. Women of non-childbearing potential may be included if surgically sterile (tubal ligation or hysterectomy) or postmenopausal with at least 2 year without spontaneous menses.
* Subject understands the study procedures and agrees to participate in the study by giving written informed consent.

Exclusion Criteria:

* Subject is under age of legal consent, male, pregnant or breastfeeding.
* Subject with a BMI ≤ 25 kg/m² or BMI ≥ 30 kg/m².
* Subject is on a diet to induce weight loss or any other treatment for obesity.
* Subject has current symptoms or a history of gastrointestinal or other significant somatic or psychiatric diseases or drug allergies.
* Subject has diabetes.
* Subject has a significant heart, lung, liver or kidney disease.
* Subject has a QT-interval > 450 ms.
* Subject has any history of a neurological disorder.
* Subject has a history of abdominal surgery. Those having undergone a simple appendectomy more than 1 year prior to the screening visit may participate.
* Subject has retinopathy.
* Subject suffers from psoriasis.
* Subject has porphyria.
* Subject shows abnormal eating behavior or has an eating disorder.
* History or current use of drugs that can affect glycaemia, gastrointestinal function, motility or sensitivity or gastric acidity.
* History or current use of centrally acting medication, including antidepressants, antipsychotics and/or benzodiazepines (in the last year before screening visit).
* Subject consumes excessive amounts of alcohol, defined as >14 units per week.
* Subject is currently (defined as within approximately 1 year of the screening visit) a regular or irregular user (including "recreational use") of any illicit drugs (including marijuana) or has a history of drug (including alcohol) abuse. Further, patient is unwilling to refrain from the use of drugs during this study.
* High caffeine intake (> 500 ml coffee daily or equivalent).
* Inability or unwillingness to perform all of the study procedures, or the subject is considered unsuitable in any way by the principal investigator.
* Recent participation (<30 days) or simultaneous participation in another clinical study.
* Subjects with lactose intolerance.
* Subjects with quinine allergy.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female volunteers have a higher chance to be more sensitive for bitter compounds because of their genetic background in comparison to males.
Enrollment: 40 (Estimated)
Dates: Start 2019-10-01 (Estimated); Primary Completion 2020-10-01 (Estimated); Study Completion 2020-10-01 (Estimated)

PRIMARY OUTCOMES:
The effect of hydroxychloroquine sulphate on hedonic food intake | 60 min after plaquenil or placebo administration
  Hedonic food intake will be assessed using a chocolate milkshake drinking task. Subjects are instructed to drink ad libitum from a chocolate milkshake until fully satiated. The milkshake will be weighted before and after the experiment and 1 g of chocolate milkshake = 1 kcal.

SECONDARY OUTCOMES:
The effect of hydroxychloroquine sulphate on gastrointestinal hormone release | First sample 10 min prior to administration. Followed by collections every 10 min after administration for a period of one hour. A final blood sample will be collected 30 min after consumption of the chocolate milkshake.
  Gastrointestinal hormone release will be measured in plasma samples collected at regular time points to assess the release of ghrelin and motilin.
The effect of hydroxychloroquine sulphate on glucose | First sample 10 min prior to administration. Followed by collections every 10 min after administration for a period of one hour. A final blood sample will be collected 30 min after consumption of the chocolate milkshake.
  Whole blood glucose levels will be measured at regular time points with a blood glucose meter.
The effect of hydroxychloroquine sulphate on appetite-related sensations | All appetite-related sensations will be scored every 10 min for a period of 110 minutes, starting 20 min before plaquenil or placebo administration and ending 90 min after administration..
  Hunger, prospective food consumption, satiety, fullness, bloating, belching, cramps and pain will be scored by the subjects on visual analog scales of 100 mm.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Tack, Principal Investigator — UZ Leuven